CLINICAL TRIAL: NCT01907204
Title: Evaluation of Inhaled Corticosteroid Treatment in Sinusitis
Brief Title: Evaluation of Inhaled Treatment in Sinusitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, G.Reychler, Docteur Gregory Reychler, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sinusitis001
Record Dates: First submitted 2013-07-12; First posted 2013-07-24 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis | interventions — Methylprednisolone; Budesonide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oral (Active Comparator): Oral drug (methylprednisolone) administration
  Interventions: Drug: methylprednisolone
- Metered dose inhaler (Experimental)
  Interventions: Drug: Budesonide
- Nebulized (Experimental)
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: methylprednisolone — Oral 32mg/8d-16mg/4d-8mg/4d
  Arms: Oral
Drug: Budesonide — Budesonide by metered dose inhaler
  Arms: Metered dose inhaler
Drug: Budesonide — Budesonide by nebulization
  Arms: Nebulized

SUMMARY:
The purpose of this study is to determine whether inhaled corticosteroid (specially nebulized) could be a good alternative to oral corticosteroid and whether they are effective in the treatment of sinusitis

ELIGIBILITY:
Inclusion Criteria:

* Nasal/Sinus polyps

Exclusion Criteria:

* Previous sinus surgery
* Age under 18y
* Use of antibiotics

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Sniffin' Sticks Test | Baseline and day 15

SECONDARY OUTCOMES:
Specific quality of life questionnaire (Snot 20) | Baseline and day 15
Retro Olfaction Test | Baseline and day 15

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Reychler, PhD, Study Director — Cliniques universitaires Saint-Luc- Université Catholique de Louvain; Philippe Rombaux, Prof PhD, Study Director — Cliniques universitaires Saint-Luc- Université Catholique de Louvain; Coralie Colbrant, PT, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain